CLINICAL TRIAL: NCT04615312
Title: Phase I Clinical Study on the Safety and Tolerability of a CDK4 / 6 Inhibitor and a MEK Inhibitor in the Treatment of Metastatic Digestive System Tumors
Brief Title: A Trail of CDK4 / 6 Inhibitor and MEK Inhibitor in the Treatment of Metastatic Digestive System Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, LiNing, Chief Physician, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRC-PANC-IIT-SHR6390-SHR7390
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Digestive System Tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- a CDK4 / 6 inhibitor and a MEK inhibitor (Experimental): Participants will receive a CDK4 / 6 inhibitor and a MEK inhibitor treatment
  Interventions: Drug: a CDK4 / 6 inhibitor and a MEK inhibitor

INTERVENTIONS:
Drug: a CDK4 / 6 inhibitor and a MEK inhibitor — Participant will receive a CDK4 / 6 inhibitor and a MEK inhibitor treatment to determine the maximum tolerated dose

SUMMARY:
This is a prospective, open, phase I clinical study to evaluate the safety and tolerability of a CDK4 / 6 inhibitor and a MEK inhibitor in the treatment of metastatic digestive system tumors

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years;
2. ECOG score ≤ 1;
3. Patients with advanced KRAS mutation or metastatic digestive system tumor confirmed by histology or cytology and imaging diagnosis;
4. According to Recist1.1, there was at least one measurable lesion;
5. The expected survival time was more than 12 weeks;

Exclusion Criteria:

1. Patients who received any anti-tumor treatment within 4 weeks before enrollment, including radiotherapy, chemotherapy, molecular targeted therapy and immunotherapy, or participated in another intervention clinical trial;
2. Previous treatment with targeted BRAF, MEK, ERK or CDK family related inhibitors;
3. The third space effusion (such as massive pleural effusion or ascites) with clinical symptoms that cannot be controlled by drainage or other methods;
4. Allergy to any test drug and its excipients, or serious allergic history, or contraindication of the test drug;
5. Have a history of immunodeficiency, including HIV positive, or other acquired, congenital immunodeficiency diseases, or a history of organ transplantation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-11-14 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose of a CDK4 / 6 inhibitor and a MEK inhibitor therapy | Up to approximately 24 months

SECONDARY OUTCOMES:
ORR | Up to approximately 24 months
  the Objective Remission Rate

CONTACTS AND LOCATIONS:
Overall Officials: Ning Li, PhD, Principal Investigator — Henan Cancer Hospital; Suxia Luo, PhD, Principal Investigator — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No